CLINICAL TRIAL: NCT01345162
Title: Randomized, Prospective Study of the Assessment, Prevention and Management of Acute Post-herniotomy Pain
Brief Title: Assessment and Prevention of Acute Post-herniotomy Pain
Acronym: PTSM04APHP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011856-23
Record Dates: First submitted 2011-04-19; First posted 2011-04-29 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Hernia
Keywords: Herniotomy
MeSH Terms: conditions — Hernia | interventions — Ketorolac Tromethamine; Ketorolac; Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketorolac (Other): Patients will be given intraoperative analgesia with Ketorolac and tramadol before the the end of surgery, then Ketorolac postoperative 10mg 1cp x 3/die, from the day of surgery for 4 days after surgery.
  Interventions: Drug: Ketorolac postoperative; Drug: intraoperative analgesia
- acetaminophene+tramadol (Other): Patients will be given intraoperative analgesia with Ketorolac and tramadol before the the end of surgery, then postoperative Patrol (acetaminophene 325mg+tramadol 37,5mg) 1cp x 3/die for 4 days after surgery.
  Interventions: Drug: postoperative Patrol; Drug: intraoperative analgesia

INTERVENTIONS:
Drug: Ketorolac postoperative — Ketorolac 10mg 1cp x 3/die
  Other Names: Toradol
  Arms: ketorolac
Drug: postoperative Patrol — acetaminophene 325mg+tramadol 37.5mg, 1cp x 3/die
  Other Names: Patrol
  Arms: acetaminophene+tramadol
Drug: intraoperative analgesia — ketorolac 30 mg iv
  Other Names: Ketorolac
Drug: intraoperative analgesia — Tramadol 100 mg if Weight over 50 kg, 50 mg if weight below 50 kg
  Other Names: Tramadol

SUMMARY:
The aim of the study is the assessment and management of Acute Post-herniotomy Pain using two different therapeutical protocols per os: ketorolac versus association of acetaminophene+tramadol.

DETAILED DESCRIPTION:
Persistent post-herniotomy pain (PPP) affects everyday activities in 5-10% of patients. Even brief intervals of acute pain can induce long-term neuronal remodeling and sensitization, chronic pain and lasting psychological distress. Chronic pain may be caused by intense acute PPP, intraoperative nerve injury and/or ongoing inflammation or mesh response with subsequence damage to nerve structures. The aim of our study is to analyze analgesic efficacy, safety and prevention of persistent postsurgical pain of two different pharmacological strategies.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years, under 80 years, scheduled for elective herniotomy
* Classification American Society of Anesthesiologists (ASA) I: without systemic disease
* Classification ASA II or III (mild systemic disease or severe systemic disease that limits the activity without invalidity).
* Patients with hernia typ 2, 3a, 3b (classification NYHUS (1993))
* Signed informed consent

Exclusion Criteria:

* ASA III, IV
* Emergency surgery
* Recovery in intensive care unit after surgery
* habitual opioid consumption
* NSADs allergy
* cognitive or mental alterations
* coagulopathy
* piastrinemia < 100.000/mm3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Cavalloro, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Matteo, Pavia, Lomabardy
  - Ospedale di Circolo e Fondazione Macchi, Varese, Lombardy

REFERENCES:
- [Derived] Bugada D, Lavand'homme P, Ambrosoli AL, Klersy C, Braschi A, Fanelli G, Saccani Jotti GM, Allegri M; SIMPAR group. Effect of postoperative analgesia on acute and persistent postherniotomy pain: a randomized study. J Clin Anesth. 2015 Dec;27(8):658-64. doi: 10.1016/j.jclinane.2015.06.008. Epub 2015 Aug 30. PMID 26329661

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac: Ketorolac 10mg
  1cp x 3/die
  postoperative analgesic treatment: 1. Ketorolac 10mg 1cp x 3/die 2. Acetaminophene 325mg+Tramadol 37,5mg 1cp x 3/die
- Acetaminophene + Tramadol: acetaminophene 325mg+tramadol 37,5mg
  1cp x 3/die
  postoperative analgesic treatment: 1. Ketorolac 10mg 1cp x 3/die 2. Acetaminophene 325mg+Tramadol 37,5mg 1cp x 3/die
Period: Overall Study
Arm/Group | Ketorolac | Acetaminophene + Tramadol
Started | 100 | 100
Completed | 98 | 96
Not Completed | 2 | 4
Not completed — Protocol Violation | 2 | 4

BASELINE CHARACTERISTICS:
Population: patients enrolled who completed the evaluations
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Acetaminophene + Tramadol | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14.6) | 56.6 (15) | 56.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 93 | 87 | 180

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Efficacy
Description: percentage of patients with NRS≥4. (NRS=numeric rating scale; o quantify pain from0=no pain to 10=worst pain possible).
  NRS≥4 is cosidered as suboptimal pain control worth to be treated with adjunctive analgesics. We therefore condidered the difference in percentage of patients experiencing not optimal pain control in the two groups to understand, if any, the difference in analgesic efficacy between the two drugs.
Time Frame: 4 days postherniotomy
Measure: Number; unit: percentage of patients with NRS≥4
Arm/Group | Ketorolac | Acetaminophene + Tramadol
Number analyzed (Participants) | 98 | 96
percentage of patients with NRS≥4 | 26.5 | 32.3

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: All adverse events (eg: PONV (postoperative nausea and vomiting), itching, dizziness, epigastralgia) are recorded.
  Assessment of any difference between the two groups.
Time Frame: 4 days postherniotoy
Reporting Status: Not Posted

3. Secondary Outcome: Difference in Recovering Daily Activity
Description: Assessment of the difference in recovering daily activity in terms of NRSm (Numeric Rate Scale at movement)
Time Frame: 4 days after surgical procedure
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of Any Connections Between the Two Therapeutical Strategies and the Recurrence of Surgical Complications
Description: Assessment of the recurrence of surgical complications. Evaluation of all the patients after 5 days by clinical evaluation. After 1 and 3 month in the patients who refer pain.
  Assessment of any difference between the two groups.
Time Frame: 4 days postherniotomy
Reporting Status: Not Posted

5. Secondary Outcome: Development of Persistent Postoperative Pain
Description: Assessment of pain prevalence and presentation of persistant postoperative pain. Evaluation of all the patients after 1 and 3 months by phone call and with clinical re-evaluation in all patients who referred pain.
Time Frame: Up to 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ketorolac | Acetaminophene + Tramadol
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/96
Other Adverse Events (participants affected / at risk) | 6/98 | 12/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=98) | Acetaminophene + Tramadol (N=96)
stipsis (Gastrointestinal disorders) | 5 (5) | 9 (9)
bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
vertigo headache parestesia (Nervous system disorders) | 2 (2) | 5 (5)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
reactive hydrocele (Renal and urinary disorders) | 1 (1) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No